CLINICAL TRIAL: NCT03249883
Title: Evaluation of a Geriatric Foot- 1M10 ADJUST Versus the Solid Ankle Cushioned Heel Foot for Low Activity Amputees
Brief Title: Comparison of Prosthetic Feet for the Geriatric Patients(CPF)
Acronym: CPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loewenstein Hospital (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0027-14-LOE
Record Dates: First submitted 2017-06-26; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Amputation
Keywords: prosthetic feet; double blind study; limited ambulators; SACH foot; prosthetic components comparison

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SACH first (Active Comparator): Will use a SACH foot for the first three weeks of prosthetic gait training , and a 1M10 foot for the second three weeks of prosthetic gait training
  Interventions: Device: SACH prosthetic foot, 1M10 prosthetic foot
- 1M10 first (Active Comparator): Will use a 1M10 foot for the first three weeks of prosthetic gait training , and a SACH foot for the second three weeks of prosthetic gait training
  Interventions: Device: SACH prosthetic foot, 1M10 prosthetic foot

INTERVENTIONS:
Device: SACH prosthetic foot, 1M10 prosthetic foot — In the SACH first group - the amputees will wear the SACH feet for three weeks and then switch to 1M10 feet for another three weeks.
  In the 1M10 first group - the amputees will wear the 1M10 feet for three weeks and then switch to SACH feet for another three weeks.

SUMMARY:
The purpose of this study is to determine whether the geriatric prosthetic foot 1M10 is superior to the classical SACH (Solid Ankle Cushion Heel) foot, when used by indoor ambulators with a transtibial amputation.

DETAILED DESCRIPTION:
Fourteen limited ambulators , unilateral trans tibial amputees, will be recruited in the orthopedic rehabilitation department in our institute. Participants will be assigned randomly to be fitted with a SACH or a 1M10 Otto Bock foot in their prosthesis.

Both types of feet will be "dressed" to look similarly. All participants will receive the same rehabilitation protocol. After three weeks all participants will be tested functionally in the "10 meter walk test" , and a "Get up and go test". The participants will answer a satisfaction questionnaire that is based on the "Prosthesis Evaluation Questionnaire" and modified according to the aims of this trial.

Pressure patterns and gait parameters will be recorded using a pressure mat. At this time the foot will be switched to the other study prosthetic foot, and the rehabilitation will commence.

At the end of three weeks wearing the new foot the same set of tests will be run again.

The investigators aim to present the difference in satisfaction and in the functional performance of the same participant wearing the two feet.

ELIGIBILITY:
Inclusion Criteria:

* unilateral transtibial amputees
* limited ambulators

Exclusion Criteria:

* do not speak Hebrew
* are not cognitively intact

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Prosthetic satisfaction Questionnaire | Measured after 3 weeks
  Hebrew satisfaction questionnaire
10 meter walk test | Measured after 3 weeks
  The participants will be asked to walk at their comfort pace 10 meters. The time of completing the task will be recorded
Get up and go test | Measured after 3 weeks
  The participants will be asked to get up from a chair walk 3 meters turn around walk back to the chair and sit down. The time of completing the task will be recorded.
Prosthetic Satisfaction Questionnaire | Measured after 6 weeks
  Hebrew satisfaction questionnaire
10 meter walk test | Measured after 6 weeks
  The participants will be asked to walk at their comfort pace 10 meters. The time of completing the task will be recorded
Get up and go test | Measured after 6 weeks
  The participants will be asked to get up from a chair walk 3 meters turn around walk back to the chair and sit down. The time of completing the task will be recorded

SECONDARY OUTCOMES:
Gait patterns | Measured after 3 weeks and
  Digital foot pressure patterns and gait parameters of the participants walking on a gait mat.
Gait patterns | Measured after 6 weeks
  Digital foot pressure patterns and gait parameters of the participants walking on a gait mat.

CONTACTS AND LOCATIONS:
Overall Officials: Hagay Amir, MD, Principal Investigator — Director of Orthopedic rehabilitation Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chitragari G, Mahler DB, Sumpio BJ, Blume PA, Sumpio BE. Prosthetic options available for the diabetic lower limb amputee. Clin Podiatr Med Surg. 2014 Jan;31(1):173-85. doi: 10.1016/j.cpm.2013.09.008. PMID 24296024
- [Result] Agrawal V, Gailey RS, Gaunaurd IA, O'Toole C, Finnieston A, Tolchin R. Comparison of four different categories of prosthetic feet during ramp ambulation in unilateral transtibial amputees. Prosthet Orthot Int. 2015 Oct;39(5):380-9. doi: 10.1177/0309364614536762. Epub 2014 Jun 12. PMID 24925671
- [Result] Bonnet X, Adde JN, Blanchard F, Gedouin-Toquet A, Eveno D. Evaluation of a new geriatric foot versus the Solid Ankle Cushion Heel foot for low-activity amputees. Prosthet Orthot Int. 2015 Apr;39(2):112-8. doi: 10.1177/0309364613515492. Epub 2014 Jan 13. PMID 24418934
- [Result] Graham LA, Fyfe NC. Prosthetic rehabilitation of amputees aged over 90 is usually successful. Disabil Rehabil. 2002 Sep 10;24(13):700-1. doi: 10.1080/09638280210142194. PMID 12296985
- [Result] Vickers DR, Palk C, McIntosh AS, Beatty KT. Elderly unilateral transtibial amputee gait on an inclined walkway: a biomechanical analysis. Gait Posture. 2008 Apr;27(3):518-29. doi: 10.1016/j.gaitpost.2007.06.008. Epub 2007 Aug 17. PMID 17707643
- [Result] Edelstein JE. Prosthetic feet. State of the Art. Phys Ther. 1988 Dec;68(12):1874-81. doi: 10.1093/ptj/68.12.1874. PMID 3057523
- [Result] Hansen A, Sam M, Childress D. The effective foot length ratio: a potential tool for characterization and eval¬uation of prosthetic feet. J Prosthet Orthot 2004; 16(2): 41-45.
- [Result] Hansen AH, Meier MR, Sessoms PH, Childress DS. The effects of prosthetic foot roll-over shape arc length on the gait of trans-tibial prosthesis users. Prosthet Orthot Int. 2006 Dec;30(3):286-99. doi: 10.1080/03093640600816982. PMID 17162519
- [Result] Arifin N, Abu Osman NA, Ali S, Wan Abas WA. The effects of prosthetic foot type and visual alteration on postural steadiness in below-knee amputees. Biomed Eng Online. 2014 Mar 5;13(1):23. doi: 10.1186/1475-925X-13-23. PMID 24597518
- [Result] Nederhand MJ, Van Asseldonk EH, van der Kooij H, Rietman HS. Dynamic Balance Control (DBC) in lower leg amputee subjects; contribution of the regulatory activity of the prosthesis side. Clin Biomech (Bristol). 2012 Jan;27(1):40-5. doi: 10.1016/j.clinbiomech.2011.07.008. Epub 2011 Sep 1. PMID 21889241
- [Result] Buckley JG, O'Driscoll D, Bennett SJ. Postural sway and active balance performance in highly active lower-limb amputees. Am J Phys Med Rehabil. 2002 Jan;81(1):13-20. doi: 10.1097/00002060-200201000-00004. PMID 11807327
- [Result] Goh JC, Solomonidis SE, Spence WD, Paul JP. Biomechanical evaluation of SACH and uniaxial feet. Prosthet Orthot Int. 1984 Dec;8(3):147-54. doi: 10.3109/03093648409146077. PMID 6522257
- [Result] Quesada PM, Pitkin M, Colvin J. Biomechanical evaluation of a prototype foot/ankle prosthesis. IEEE Trans Rehabil Eng. 2000 Mar;8(1):156-9. doi: 10.1109/86.830960. PMID 10779119